CLINICAL TRIAL: NCT03996109
Title: Living Green and Healthy for Teens (LiGHT) - a Randomized Trial Evaluating Behaviour Change Using a Gamified Healthy Living App for Youth and Their Families
Brief Title: Living Green and Healthy for Teens
Acronym: LiGHT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Childhood Obesity Foundation (Other); University of British Columbia (Other); Ayogo Health Inc. (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LiGHT
Record Dates: First submitted 2019-06-19; First posted 2019-06-24 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Healthy Lifestyle; Adolescent Behavior
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aim2Be (Experimental): Youth-parent dyads randomized to Aim2Be
  Interventions: Behavioral: Aim2Be smartphone app system
- BnLt (Active Comparator): Youth-parent dyads randomized to BnLt
  Interventions: Behavioral: BnLt smartphone app

INTERVENTIONS:
Behavioral: Aim2Be smartphone app system — Youth-parent dyads will receive the LiGHT program (addressing healthy eating, physical activity, screen time and sleep) via the Aim2Be smartphone app for 6 months. It provides personalization beginning with creation of an avatar and identifying user motivations, offers progressive goal-setting considering readiness, sub-tasks, milestones, self-monitoring tools with feedback and positive reinforcement. It applies behaviour change techniques, provides a knowledge centre, simulation narratives to enable decision making, and separate social exchange platforms for parents and youth to share ideas and challenges with peers. A Virtual Coach has been programmed using motivational interviewing theory. Gamification includes elements of choice, challenge, uncertainty, discovery, and kudos for achieving outcomes in the process of developing motivations, skills and mastery.
  Arms: Aim2Be
Behavioral: BnLt smartphone app — Youth-parent dyads will receive a simple app called BnLt for 6 months. It provides web-links to external websites that provide information and tips on healthy eating and activity, including the Canada Food Guide, Canadian Society of Exercise Physiology recommendations for physical activity, screen time and sleep for youth, and other resources.
  Arms: BnLt

SUMMARY:
This is a two-group parallel randomized controlled trial testing whether a gamified healthy living smartphone app for youth aged 10-16 representative of the Canadian population and one of their parents is more effective at improving a composite of health behaviours (diet, physical activity, sleep and screen time) than a simple app providing links to healthy living websites.

DETAILED DESCRIPTION:
Living Green and Healthy for Teens (LiGHT) is a Canadian smartphone app-based program that combines health promotion (healthy eating, active living, screen time and sleep) with additional novel motivators such as environmental stewardship (e.g. reduce prepackaged foods, walk rather than drive) and cost-savings (e.g., eat at home rather than restaurants), that may further increase the likelihood of behaviour change.

The primary aim of the trial is to determine, among youth aged 10-16 years, if randomization of their family to the use of the interactive gamified Living Green and Healthy for Teens (LiGHT) app over a 6 month period, compared to a control app, increases the number of healthy active living behaviours engaged in by youth. Additional outcomes will include youth anthropometrics, diet quality, fitness, quality of life, and parental health behaviours and cardiovascular risk.

Using a multi-centre randomized, parallel, controlled single-blind design, 376 eligible youth-parent dyads stratified by youth (gender, and age <13.5/≥13.5y) will be allocated 1:1 to receive intervention or control apps that provide information and tips on healthy eating and activity in different ways. Participants will be followed for 1 year, with the primary outcome assessed at 6 months.

Participants will be recruited from the community in Hamilton, Ontario, and Surrey, British Columbia, Canada. The target population is the general population of youth and their families. Therefore, entry criteria will be broad. Youth aged 10-16 years of age who identify a need or potential to improve health behaviours will be included if one parent is willing to attend all study visits and use the app, there is at least one internet enabled device in the household, and there are no contraindications to healthy eating and activity, and no family member is participating in a weight management program or other clinical trial.

Participants will be blinded to treatment group. Both apps have appealing interfaces, and both provide information, tips and interactivity (though to different degrees). Every effort will be made to keep research staff who help participants with the app separate from staff who collect data, and the latter will be trained to avoid discussing the intervention.

Evaluations at baseline, 3 months and 6 months by virtual or in-person appointments will include a youth questionnaire including questions about food intake , screen time, physical activity, health related quality of life, and resilience, and measurement of height, weight, and fitness using a push-up test and standing long jump test. Participants completing in-person visits will also complete the following: body fat percentage using bioelectrical impedance assessment, blood pressure, hand grip strength using a dynamometer, and cardiorespiratory fitness using a step test. Youth participants will also provide a urine sample and wear an accelerometer for 7 days. Parents will complete a questionnaire including questions about sociodemographics, their own food intake, screentime, physical activity, parental role modelling and logistic support. Parents will also complete the non-laboratory based INTERHEART risk score questionnaire and have their waist and hip circumference measured. Participants and parents will complete questionnaires about youth experience of online bullying and access to undesirable online content. 12 months after randomization, participants and parents may be invited to complete the same study questionnaires online.

This trial will demonstrate whether use of a rigorously-designed, evidence-based, user-friendly app is able to help families with teenagers improve health behaviours of youth and have any early impact on CV risk factors. Conducting an RCT in the context of the full range of youth in the community has the potential to inform population-scale implementation as a public health tool for sustainable obesity prevention across Canada.

ELIGIBILITY:
Inclusion Criteria:

1. Living in a home setting with at least one smartphone or tablet and internet access in the household, and
2. One parent or guardian (the "primary parent") who is able to attend all study visits.
3. Youth or parent identifying a need or potential to improve health behaviours

Exclusion Criteria:

1. Inability of the youth and/or primary parent to read English at a grade 5 level
2. A health condition in the youth that precludes eating a variety of foods or engaging in physical activity
3. Current participation of any family member in a weight management program
4. Current participation in another clinical trial
5. Current or prior participation of another member of the household/family in this trial

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2021-12-11 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Healthy living behaviours | 6 months
  Number of behaviours engaged in by youth of the following 7 behaviours: a) ≥60 minutes of MVPA daily, b) ≤2 hours of recreational screen time daily, c) 9-11 hours (for those ≤13 years) and 8-10 hours (for those ≥14 years) of nightly sleep, d) ≥5 fruit and vegetable servings per day, e) ≤2 sugary beverages per week, f) breakfast consumption 7 days per week, and g) eating out or ordering in <1 time per week.

SECONDARY OUTCOMES:
BMI Z-score | 6 months
  Age, and sex specific body mass index Z-scores based on WHO norms
MVPA | 6 months, 1 year
  Average daily minutes of moderate to vigorous physical activity measured by accelerometry over 1 week
Diet quality biomarker | 6 months
  Diet quality assessed by urine sodium-to-potassium concentration ratio

OTHER OUTCOMES:
Change in number of health behaviours | 6 months, (1 year exploratory)
  Change from baseline in the number of the 7 measured health behaviours over time
Cardiorespiratory fitness | 6 months
  The modified Canadian Aerobic Fitness Test step test (Score range 0-4 with higher scores indicating better fitness)
Health related quality of life | 6 months, (1 year exploratory)
  Kidscreen-27 Health-Related Quality of Life Questionnaire for Children and Adolescents - Total Score and Subscales(Physical Well-Being, Psychological Well-Being, Autonomy & Parents, Peers & Social Support, and School Environment) - Total and subscales transformed to T scores with mean 50 and standard deviation 10 with higher scores indicating better quality of life
Child and Youth Resilience Measure-12 | 6 months, (1 year exploratory)
  The Child and Youth Resilience Measure (CYRM) is a questionnaire assessing the resources (individual, relational, communal and cultural) available to individuals that may bolster their resilience. (Score range 12-36 with higher scores indicating better resilience)
Parental support of healthy eating and physical activity | 6 months, (1 year exploratory)
  Survey questions to asses parental role-modelling and logistic support of their youth's eating and activity behaviours
Changes in parental diet | 6 months, (1 year exploratory)
  Changes in parental mean frequency of intake of fruits & vegetables, sugary drinks, eating breakfast and restaurant meals from baseline
Changes in parental physical activity | 6 months, (1 year exploratory)
  Changes in parental metabolic equivalent-minutes (MET-mins) from the International Physical Activity Questionnaire (Score range 0-19278, with higher scores indicating greater physical activity)
Parental cardiovascular risk | 6 months, (1 year exploratory)
  Parental non-laboratory based Interheart modifiable cardiovascular risk score, including questions about diabetes, hypertension, smoking, stress, family history, diet and physical activity (Score range 0-48, with higher scores indicating greater cardiovascular risk)

CONTACTS AND LOCATIONS:
Overall Officials: Zubin Punthakee, MD, MSc, Principal Investigator — Population Health Research Institute
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada